CLINICAL TRIAL: NCT05963022
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of Tirzepatide Monotherapy Compared With Placebo in Chinese Participants With Type 2 Diabetes
Brief Title: A Study of Tirzepatide (LY3298176) in Chinese Participants With Type 2 Diabetes (SURPASS-CN-MONO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18746; I8F-MC-GPIU (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 5 Milligram (mg) Tirzepatide (Experimental): Participants received 5 mg of tirzepatide administered as subcutaneous (SC) injection via a single-dose pen (SDP) once weekly (QW) for 40 weeks.
  The starting dose of tirzepatide was 2.5 mg QW, which increased by 2.5 mg every 4 weeks until the maintenance dose of 5 mg was reached.
  Interventions: Drug: Tirzepatide
- 10 mg Tirzepatide (Experimental): Participants received 10 mg of tirzepatide administered as SC injection via a SDP QW for 40 weeks.
  The starting dose of tirzepatide was 2.5 mg QW, which increased by 2.5 mg every 4 weeks (2.5 mg to 5 mg to 7.5 mg to 10 mg) until the maintenance dose of 10 mg was reached.
  Interventions: Drug: Tirzepatide
- 15 mg Tirzepatide (Experimental): Participants received 15 mg of tirzepatide administered as SC injection via a SDP QW for 40 weeks.
  The starting dose of tirzepatide was 2.5 mg QW, which increased by 2.5 mg every 4 weeks (2.5 mg to 5 mg to 7.5 mg to 10 mg to 12.5 mg to 15 mg) until the maintenance dose of 15 mg was reached.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants received tirzepatide matched placebo administered as SC injection via a SDP QW for 40 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 10 mg Tirzepatide; 15 mg Tirzepatide; 5 Milligram (mg) Tirzepatide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to investigate the efficacy and safety of Tirzepatide monotherapy in Chinese participants with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes
* Have HbA1c ≥7.0% (≥53 mmol/mol) to ≤9.5% (≤80 mmol/mol) despite diet and exercise treatment
* Are of stable weight 5%) during the 90 days preceding screening and agree not to initiate a diet and/or exercise program during the study with the intent of reducing body weight other than the lifestyle and dietary measures for diabetes treatment
* Have Body Mass Index (BMI) ≥23.0 kilogram per square meter (kg/m²)

Exclusion Criteria:

* Have Type 1 Diabetes
* Have a history of chronic or acute pancreatitis any time prior to study entry
* Are currently receiving treatment for diabetic retinopathy and/or macular edema
* Have a history of ketoacidosis or hyperosmolar state/coma
* Have a history of New York Heart Association Functional Classification IV congestive heart failure (CHF)
* Have acute or chronic hepatitis including a history of autoimmune hepatitis
* Use of insulin 1-year preceding screening and between screening and baseline; use of any antihyperglycemic medication 90 days preceding screening and between screening and baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (28):
- China (28):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Shunde Hospital of Southern Medical Univesity, Foshan, Guangdong
  - Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - Zunyi First People's Hospital, Zunyi, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Yichang Central People's Hospital, Yichang, Hubei
  - The First People's Hospital of Changde City, Changde, Hunan
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing Medical University - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Dalian University - The Affiliated Zhongshan Hospital, Dalian, Liaoning
  - Dalian Municipal Central Hospital Affiliated of Dalian Medical University, Dalian, Liaoning
  - Panjin Liaoyou Baoshihua Hospital, Liaoyou, Liaoning
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Pudong New Area People's Hospital Shanghai, Shanghai, Shanghai Municipality
  - Jiading District Central Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Huzhou Central Hospital, Huzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5 Milligram (mg) Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Started | 52 | 51 | 52 | 51
Received at Least One Dose of Study Drug | 52 | 51 | 52 | 51
Completed | 52 | 46 | 48 | 47
Not Completed | 0 | 5 | 4 | 4
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 3 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Subject Required long-term Initiation of Rescue Antihyperglycemic Medication | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 5 mg Tirzepatide: Participants received 5 mg of tirzepatide administered as SC injection via a SDP QW for 40 weeks.
  The starting dose of tirzepatide was 2.5 mg QW, which increased by 2.5 mg every 4 weeks until the maintenance dose of 5 mg was reached
- Total: Total of all reporting groups
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo | Total
Number analyzed (Participants) | 52 | 51 | 52 | 51 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.30 (11.37) | 50.70 (10.79) | 50.60 (12.11) | 47.60 (11.56) | 48.80 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 25 | 22 | 90
  Male | 29 | 31 | 27 | 29 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 52 | 51 | 52 | 51 | 206
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 52 | 51 | 52 | 51 | 206
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 52 | 51 | 52 | 51 | 206
Percentage of Hemoglobin A1c (HbA1c) at Baseline [Mean (Standard Deviation); unit: Percentage of HbA1c] | 8.07 (0.77) | 8.13 (0.78) | 7.97 (0.81) | 7.92 (0.67) | 8.02 (0.76)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least squares (LS) mean was calculated using ANCOVA model with Baseline + Prior Antihyperglycemic Use + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, Week 40
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline value at the specified time point for this outcome, regardless of adherence to study intervention or initiation of rescue antihyperglycemic medication.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 52 | 44 | 48 | 47
percentage of HbA1c | -2.19 (0.121) | -1.75 (0.131) | -2.03 (0.124) | -0.77 (0.126)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -1.42, 95% CI 2-sided [-1.76 to -1.07]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.98, 95% CI 2-sided [-1.34 to -0.63]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -1.26, 95% CI 2-sided [-1.61 to -0.92]

2. Secondary Outcome: Percentage of Participants With HbA1c Target Values of <7.0% (<53 Millimole/Mole [mmol/Mol])
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. The percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, multiplied by 100. Percentage of participants with HbA1c <7.0% (<53 mmol/mol) is reported here.
Time Frame: Week 40
Population: All randomized participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 52 | 44 | 48 | 47
percentage of participants | 90.38 | 86.36 | 83.33 | 38.30
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 17.04, 95% CI 2-sided [5.62 to 51.73]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.51, 95% CI 2-sided [2.77 to 20.37]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.24, 95% CI 2-sided [2.74 to 19.14]

3. Secondary Outcome: Change From Baseline in Fasting Serum Glucose
Description: LS mean was calculated using ANCOVA model with Baseline + Prior Antihyperglycemic Use + Baseline HbA1c Group (<=8.5%, >8.5%) + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligram per deciliter (mg/dL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 51 | 46 | 48 | 49
milligram per deciliter (mg/dL) | -55.0 (3.00) | -54.8 (3.16) | -55.4 (3.06) | -30.2 (3.07)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -24.8, 95% CI 2-sided [-33.3 to -16.3]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -24.6, 95% CI 2-sided [-33.2 to -15.9]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -25.2, 95% CI 2-sided [-33.7 to -16.7]

4. Secondary Outcome: Percentage of Participants With HbA1c Target Values of ≤6.5% (≤48 mmol/Mol)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. The percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, multiplied by 100. Percentage of participants with HbA1c ≤6.5% (≤48 mmol/Mol) is reported here.
Time Frame: Week 40
Population: All randomized participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 52 | 44 | 48 | 47
percentage of participants | 88.46 | 75.00 | 81.25 | 23.40
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 25.61, 95% CI 2-sided [8.70 to 75.36]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.25, 95% CI 2-sided [2.88 to 18.25]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 10.95, 95% CI 2-sided [4.23 to 28.34]

5. Secondary Outcome: Change From Baseline in Body Weight
Description: as for outcome 3
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 52 | 46 | 48 | 49
kilograms (kg) | -6.1 (0.68) | -5.5 (0.71) | -8.7 (0.69) | -1.3 (0.70)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -4.8, 95% CI 2-sided [-6.7 to -2.9]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -4.2, 95% CI 2-sided [-6.2 to -2.3]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -7.3, 95% CI 2-sided [-9.3 to -5.4]

6. Secondary Outcome: Percentage of Participants With HbA1c Target Values of <5.7% (<39 mmol/Mol)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. The percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, multiplied by 100. Percentage of participants with HbA1c <5.7% (<39 mmol/mol) is reported here.
Time Frame: Week 40
Population: All randomized participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 52 | 44 | 48 | 47
percentage of participants | 40.38 | 34.09 | 56.25 | 0
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 76.62, 95% CI 2-sided [4.40 to 1333.29]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 49.36, 95% CI 2-sided [2.80 to 868.67]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 118.22, 95% CI 2-sided [6.80 to 2055.04]

7. Secondary Outcome: Change From Baseline in Daily Average 7-Point Self-Monitored Blood Glucose Profiles (SMBG)
Description: The SMBG data were collected at the following 7 time points: Morning Premeal - Fasting, Morning 2-hour Post meal, Midday Premeal, Midday 2-hour Post meal, Evening Premeal, Evening 2-hour Post meal and Bedtime. The daily average was calculated as the average of the 7 blood glucose values collected on a particular day. LS Mean was calculated using mixed model repeated measures (MMRM) for post-baseline measures: Variable = Baseline + Baseline HbA1c (<=8.5%, >8.5%) + Prior Antihyperglycemic Use + Treatment + Time + Treatment*Time(Type III sum of squares). Variance-Covariance structure (Change from Baseline) = Unstructured.
Time Frame: Baseline, Week 40
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline value at the specified time point for this outcome regardless of adherence to study drug or initiation of rescue antihyperglycemic medication.
Measure: Least Squares Mean (Standard Error); unit: milligram per deciliter (mg/dL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 51 | 45 | 43 | 27
milligram per deciliter (mg/dL) | -78.4 (3.959) | -78.3 (4.185) | -80.8 (4.186) | -33.9 (5.223)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -44.5, 95% CI 2-sided [-57.5 to -31.5]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -44.3, 95% CI 2-sided [-57.6 to -31.1]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -46.9, 95% CI 2-sided [-60.1 to -33.7]

8. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss of ≥5%
Description: Percentage of Participants who Achieved Weight Loss ≥5% is reported here.
Time Frame: Week 40
Population: All randomized participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 51 | 45 | 43 | 27
percentage of participants | 54.90 | 66.67 | 88.37 | 7.41
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 18.19, 95% CI 2-sided [5.27 to 62.73]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 30.96, 95% CI 2-sided [8.87 to 108.05]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 73.42, 95% CI 2-sided [19.36 to 278.40]

9. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss of ≥10%
Description: Percentage of Participants who Achieved Weight Loss ≥10% is reported here.
Time Frame: Week 40
Population: All randomized participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 51 | 45 | 43 | 27
percentage of participants | 27.45 | 33.33 | 58.14 | 0
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.011, Regression, Logistic; Odds Ratio (OR) = 39.04, 95% CI 2-sided [2.29 to 664.36]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 56.34, 95% CI 2-sided [3.34 to 949.59]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 127.52, 95% CI 2-sided [7.58 to 2145.42]

10. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss of ≥15%
Description: Percentage of Participants who Achieved Weight Loss ≥15% is reported here.
Time Frame: Week 40
Population: All randomized participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 51 | 45 | 43 | 27
percentage of participants | 9.80 | 13.33 | 37.21 | 0
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.077, Regression, Logistic; Odds Ratio (OR) = 13.86, 95% CI 2-sided [0.75 to 254.78]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.062, Regression, Logistic; Odds Ratio (OR) = 15.65, 95% CI 2-sided [0.87 to 281.74]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 66.69, 95% CI 2-sided [3.90 to 1140.13]

ADVERSE EVENTS:
Time Frame: Baseline up to week 44
Description: All randomized participants who received at least one dose of study drug regardless of adherence to study drug or initiation of rescue antihyperglycemic medication. Based on the planned safety analysis, adverse events were collected per the treatment regimen, irrespective of each dose level. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/51 | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 5/52 | 6/51 | 3/52 | 5/51
Other Adverse Events (participants affected / at risk) | 41/52 | 44/51 | 45/52 | 36/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide (N=52) | 10 mg Tirzepatide (N=51) | 15 mg Tirzepatide (N=52) | Placebo (N=51)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/23 (0) | 1/20 (1) | 0/25 (0) | 0/22 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1/23 (1) | 0/20 (0) | 0/25 (0) | 0/22 (0)
Nasal cavity mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide (N=52) | 10 mg Tirzepatide (N=51) | 15 mg Tirzepatide (N=52) | Placebo (N=51)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 8 (16) | 6 (9) | 6 (6) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (5) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 12 (19) | 12 (21) | 15 (41) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (2) | 4 (13) | 3 (21) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (9) | 11 (19) | 14 (34) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 3 (4) | 3 (4) | 5 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (5) | 10 (17) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (6) | 3 (3) | 1 (1)
Injection site reaction (General disorders) | 2 (7) | 2 (32) | 5 (27) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 3 (4) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 5 (6) | 1 (1) | 1 (1) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 11 (14) | 9 (12) | 9 (13) | 10 (17)
Vaginal infection (Infections and infestations) | 0/23 (0) | 1/20 (1) | 0/25 (0) | 2/22 (2)
Amylase increased (Investigations) | 2 (2) | 2 (2) | 5 (6) | 0 (0)
Lipase increased (Investigations) | 4 (4) | 2 (4) | 4 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 15 (18) | 13 (21) | 14 (19) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 2 (2) | 17 (17)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 0 (0) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 4 (4) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 3 (3) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1/23 (1) | 1/20 (1) | 0/25 (0) | 1/22 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 0/23 (0) | 1/20 (1) | 0/25 (0) | 0/22 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 4 (4) | 0 (0) | 5 (5)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT05963022/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT05963022/SAP_001.pdf